CLINICAL TRIAL: NCT03790189
Title: Subchondral and Intra-articular Application of Bone Marrow Concentrate as a Treatment Strategy for Knee Unicompartmental Osteoarthritis (OA): a Pilot Trial
Brief Title: Subchondral and Intra-articular Application of Bone Marrow Concentrate for Knee Unicompartmental OA
Acronym: MarrowMule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 172797
Record Dates: First submitted 2018-12-22; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis, Knee; Cartilage Degeneration
Keywords: knee; unicompartmental osteoarthritis; injection; subchondroplasty; bone marrow concentrate; mesenchymal stem cells
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Marrow Concentrate (Experimental): Bone Marrow concentrate will be injected intra-articularly and at the bone-cartilage interface both in the tibia and femur of patients affected by unicompartmental knee osteoarthritis
  Interventions: Biological: Subchondral and intra-articular injection of BMC

INTERVENTIONS:
Biological: Subchondral and intra-articular injection of BMC — Bone Marrow concentrate will be injected intra-articularly and at the bone-cartilage interface both in the tibia and femur of patients affected by unicompartmental knee osteoarthritis

SUMMARY:
Unicompartmental knee osteoarthritis (OA) is a common finding especially in patients with lower limb malalignment and previous meniscectomy. Among the various treatment options, in recent years there has been an increasing attention towards the use of biologic agents, such as platelet rich plasma and mesenchymal stem cells, as intra-articular injective approaches to relieve pain and restore joint function. Anyway, the sole intra-articular administration of these agents may not lead to satisfactory outcome in a relevant percentage of patients. In fact, unicompartmental osteoarthritis is not only characterized by degeneration of the articular cartilage, but also by pathologic changes in the subchondral bone, both at the tibial plateaux and in the femoral condyle. Magnetic resonance imaging reveals, in many cases, alterations of the subchondral tissue known as "bone marrow edema", which is a sign of bone overload and play a significant role in the progression of unicompartmental OA and is responsible of OA-related symptoms. Therefore, concurrent treatment of both the subchondral bone damage and intra-articular degeneration could led to better outcome for patients affected by unicompartmental OA: the aim of the present pilot trial is to assess the safety and describe the clinical outcome following concurrent intra-articular and subchondral bone application of Bone Marrow Concentrate (BMC). BMC is an autologous product rich in mesenchymal stem cells, which have immuno-modulatory and throfic properties and are able to restore the joint homeostasis by reducing the inflammatory distress traditionally associated to OA.

BMC will be collected directly in the operating room from the anterior iliac crest or the tibia by using the MARROW CELLUTION kit (Geistlich, Switzerland), which allows to obtain BMC without the need of centrifugation processes. Approximately 9-10 ml of BMC will be harvested: 6 ml will be injected, under fluoroscopic guidance, in the tibial emiplateaux (approx 3 ml) and in the femoral condyle (approx 3 ml) presenting MRI evidence of bone marrow edema. The remaining amount of BMC will be administered intra-articularly to address articular tissues (cartilage, menisci and synovium). Twenty-five patients affected by unicompartmental knee OA will be included in the present pilot trial and treated in a "Day-Surgery" regimen. They will be followed up at 3, 6, and 12 months' after treatment by clinical questionnaires and radiographic evaluations (x-rays at 6 and 12 months, MRI at 12 months' f-up). Any intra-op and post-op adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* chronic symptomatic (at least 6 months) medial or lateral unicompartmental OA of the knee, with Kellgren-Lawrence Score evaluated at x-rays= 2 or 3;
* MRI evidence of "bone marrow edema" affecting the subchondral bone of the tibial emiplateaux and femoral condyle;
* failure of previous conservative treatments in the same knee (e.g: pharmacological therapy, physiotherapy, previous intra-articular injections, etc..);
* willingness to participate in the trial, including all follow-up visits and radiographic examinations.

Exclusion Criteria:

* medial or lateral unicompartmental OA with Kellgren-Lawrence score= 1 or 4 (i.e. early osteoarthritis or end-stage osteoarthritis);
* no MRI evidence of bone marrow edema in the affected knee compartment;
* concurrent rheumatic or other immunological diseases;
* concurrent malignancies;
* bilateral symptomatic knee OA;
* concurrent patello-femoral OA;
* BMI>35
* any surgical treatment in the index knee within 12 months from the screening visit.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in IKDC (International Knee Documentation Committee) subjective score | baseline vs 12 months' follow-up
  IKDC subjective score is a validated clinical questionnaire (available also in Italian) designed to assess the functional status of the knee by a series of 10 items. The IKDC subjective score assess the overall function of the knee as subjectively evaluated by the patient who needs to answer a series of questions concerning symptoms and his/her activity level. It ranges from 0 to 100 points, with higher values representing a better knee status.

SECONDARY OUTCOMES:
Variation in KOOS (Knee Injury and Osteoarthritis Outcome) Score | baseline vs 12 months' follow-up
  KOOS score is a validated clinical questionnaire (available also in Italian) designed to assess the functional status of the knee by a series of 42 items. KOOS score consists of five sub-scales (Pain, Symptoms, Activity of Daily life, Sport, Quality of Life). The total score is obtained by summing the score of each sub-scale (max 21 point for Pain, 17 points for Symptoms, 41 points for Activity of daily life, 12 points for Sport, 9 points for Quality of Life). The total score's range is 0-100 and higher values represents better knee status.
VAS (Visual Analogue Scale) for pain | baseline vs 12 months' after treatment
  Visual Analogue Scale to evaluate average knee pain during daily life. Range is from 0 to 100 and higher values represent higher pain perceived by the patient.
MRI (Magnetic Resonance Imaging) Changes in subchondral bone edema and cartilage status from basal to 12 months' follow-up | baseline vs 12 months' follow-up
  MRI of the index knee will be performed to assess if the bone marrow concentrate was able to produce any effect on the subchondral bone edema and/or articular cartilage. To this purpose, the WORMS (Whole Organ Magnetic Resonance Imaging Score) will be adopted. This score allows to evaluate: 1) the amount of bone marrow edema (0-3 scale based on the extension of the bone marrow edema in the anatomical region considered, with higher value representing bigger bone marrow edema); 2) the cartilage damage (0 to 6 scale with higher values representing worse cartilage status)

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — Istituto Clinico Humanitas, Rozzano, Italy; Berardo Di Matteo, MD, Study Director — Istituto Clinico Humanitas, Rozzano, Italy
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez M, Delgado D, Sanchez P, Muinos-Lopez E, Paiva B, Granero-Molto F, Prosper F, Pompei O, Perez JC, Azofra J, Padilla S, Fiz N. Combination of Intra-Articular and Intraosseous Injections of Platelet Rich Plasma for Severe Knee Osteoarthritis: A Pilot Study. Biomed Res Int. 2016;2016:4868613. doi: 10.1155/2016/4868613. Epub 2016 Jul 4. PMID 27462609
- [Background] Kwan Tat S, Lajeunesse D, Pelletier JP, Martel-Pelletier J. Targeting subchondral bone for treating osteoarthritis: what is the evidence? Best Pract Res Clin Rheumatol. 2010 Feb;24(1):51-70. doi: 10.1016/j.berh.2009.08.004. PMID 20129200
- [Background] Dray A, Read SJ. Arthritis and pain. Future targets to control osteoarthritis pain. Arthritis Res Ther. 2007;9(3):212. doi: 10.1186/ar2178. PMID 17561993
- [Background] Pan J, Wang B, Li W, Zhou X, Scherr T, Yang Y, Price C, Wang L. Elevated cross-talk between subchondral bone and cartilage in osteoarthritic joints. Bone. 2012 Aug;51(2):212-7. doi: 10.1016/j.bone.2011.11.030. Epub 2011 Dec 16. PMID 22197997
- [Background] Sanchez M, Fiz N, Guadilla J, Padilla S, Anitua E, Sanchez P, Delgado D. Intraosseous infiltration of platelet-rich plasma for severe knee osteoarthritis. Arthrosc Tech. 2014 Dec 15;3(6):e713-7. doi: 10.1016/j.eats.2014.09.006. eCollection 2014 Dec. PMID 25685680
- [Background] Pretzel D, Linss S, Rochler S, Endres M, Kaps C, Alsalameh S, Kinne RW. Relative percentage and zonal distribution of mesenchymal progenitor cells in human osteoarthritic and normal cartilage. Arthritis Res Ther. 2011 Apr 15;13(2):R64. doi: 10.1186/ar3320. PMID 21496249
- [Background] Hernigou P, Auregan JC, Dubory A, Flouzat-Lachaniette CH, Chevallier N, Rouard H. Subchondral stem cell therapy versus contralateral total knee arthroplasty for osteoarthritis following secondary osteonecrosis of the knee. Int Orthop. 2018 Nov;42(11):2563-2571. doi: 10.1007/s00264-018-3916-9. Epub 2018 Mar 27. PMID 29589086